CLINICAL TRIAL: NCT01330641
Title: Accuracy of Needle Placement Into The Subacromial Space of The Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Richard A. Marder MD, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200816140
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Rotator Cuff Tendonitis
Keywords: Tendonitis; Rotator Cuff; Shoulder; Injection
MeSH Terms: conditions — Rotator Cuff Injuries; Tendinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Anterior injection Route (Active Comparator): Group of patients injected with medication using the anterior route
  Interventions: Procedure: Injection of Subacromial Bursa
- Posterior Injection (Active Comparator): Group of patients receiving injection through a posterior route
  Interventions: Procedure: Injection of Subacromial Bursa
- Lateral Injection (Active Comparator): Group of patients receiving subacromial injection through a lateral route
  Interventions: Procedure: Injection of Subacromial Bursa

INTERVENTIONS:
Procedure: Injection of Subacromial Bursa — Injection of steroid and anesthetic to relieve pain

SUMMARY:
This study attempts to determine the most accurate route for injection of the subacromial bursa in patients with rotator cuff tendonitis. Typically, in medical practice, one of the routes of injection is used. It has not been determined if one route is superior, or if all routes are equal in delivering medication into the subacromial bursa, which sits on top of the rotator cuff tendons.

DETAILED DESCRIPTION:
Patients with a diagnosis of rotator cuff tendonitis, having failed other non-operative measures, are offered an injection of steroid and local anesthetic to relieve their pain. This is standard treatment. In this study, patients are prospectively randomized to receive their injection by one of the three commonly used routes: anterior, posterior, or lateral. Accuracy of the injection is determined by including a small amount of contrast dye in the injection which will make the injection visible on post-injection radiographs.

ELIGIBILITY:
Inclusion Criteria:

* rotator cuff tendinitis

Exclusion Criteria:

* diabetes
* allergy to contrast dye
* renal disease
* pregnancy
* frozen shoulder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Radiographic e Radiographic Evidence of Successful Subacromial Injection | One-hour post injection
  After injection of the subacromial bursa, all patients had two view radiographs performed within one hour to assess the accuracy of the injections

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Marder, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Department of Orthopaedic Surgery, Sacramento, California, United States